CLINICAL TRIAL: NCT06419621
Title: A Multicenter, Randomized, Double-blind Phase III Study of PM8002 or Placebo in Combination With Nab-Paclitaxel as First-line Treatment in Inoperable Locally Advanced/Metastatic Triple-negative Breast Cancer(TNBC)
Brief Title: PM8002 or Placebo Plus Nab-Paclitaxel as First-line Treatment in Inoperable Locally Advanced/Metastatic TNBC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PM8002-C013C-TNBC-R
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Triple Negative Breast Cancer(TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PM8002 Plus Nab-Paclitaxel (Experimental): Patients will receive both PM8002 and Nab-Paclitaxel.
  Interventions: Drug: PM8002; Drug: Nab-Paclitaxel
- Placebo Plus Nab-Paclitaxel (Placebo Comparator): Patients will receive both Placebo and Nab-Paclitaxel.
  Interventions: Drug: Nab-Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: PM8002 — PM8002 20 mg/kg via intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle
  Arms: PM8002 Plus Nab-Paclitaxel
Drug: Nab-Paclitaxel — Nab-Paclitaxel 100mg/m2 via IV infusion on Days 1, 8, and 15 of each 28-day cycle
Drug: Placebo — Placebo 20 mg/kg via IV infusion on Days 1 and 15 of each 28-day cycle
  Arms: Placebo Plus Nab-Paclitaxel

SUMMARY:
This multicenter, randomized, double-blind study will evaluate the safety and efficacy of PM8002 in combination with Nab-Paclitaxel compared with placebo combined with Nab-Paclitaxel as first-line treatment in inoperable locally advanced/metastatic triple-negative breast cancer(TNBC)

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willing to provide written informed consent and to comply with scheduled visits and study procedures;
* Female, aged 18 to 70 years (inclusive);
* Histologically confirmed unresectable locally advanced or metastatic breast cancer with negative status for ER, PR, and HER-2. Testing results for all three markers conducted within 24 months prior to the initiation of the study by a local facility accredited by clinical research center are acceptable. If deemed necessary by the investigator during screening, subjects may provide additional biopsy to confirm the latest pathological;
* Subjects who have not received prior systemic treatment（except endocrine therapy） for advanced breast cancer are eligible for the study. Subjects who have received Taxane-based chemotherapy during the neoadjuvant and/or adjuvant treatment phase are eligible, as long as the occurrence of relapse or metastasis is at least 12 months after the end of treatment;
* Performance status as assessed by the Eastern Cooperative Oncology Group (ECOG) is 0-1;
* Life expectancy of 12 weeks or more;
* According to RECIST 1.1, the subject has at least 1 measurable lesion as the targeted lesion (the only bone metastasis or the only central nervous system metastasis should not be considered as a measurable lesion. A measurable lesion located at the previously irradiated radiation field or other local treatment area should not be selected as targeted lesion, unless the lesion shows unequivocal radiographic progression).

Exclusion Criteria:

* Previous treatment with immune checkpoint agonists (such as CD137 agonists) or immune checkpoint inhibitors (such as CTLA-4, PD-1, PD-L1, LAG3 monoclonal antibody, etc.) or anti-vascular endothelial growth factor (VEGF) target drugs;
* Has uncontrolled or symptomatic brain or spine cord metastases;
* Those who have had other active malignant tumors within 5 years prior to the study treatment, except for those that can be treated locally and have been cured ;
* Poorly controlled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg);
* With a history of hypertensive crisis or hypertensive encephalopathy;
* With a history of abdominal fistula, tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess within the last 6 months prior to the start of the study treatment;
* Adverse events resulting from prior anti-tumor therapies should be assessed and graded according to the CTCAE 5.0 criteria, subjects whose AEs have not returned to Grade 1 or below;
* Has uncontrollable pleural, pericardial, or abdominal effusions;
* Has received allogeneic hematopoietic stem cell transplantation or organ transplantation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) assessed by Blinded Independent Review Committee (BIRC) | Up to approximately 37 months from first patient in
  Progression-free survival is defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) based on assessments by Blinded Independent Review Committee (BIRC) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Overall Survival (OS) | Up to approximately 37 months from first patient in
  Overall survival is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis are censored at the date of the last follow-up.

SECONDARY OUTCOMES:
PFS assessed by investigator | Up to approximately 37 months from first patient in
  Progression-free survival is defined as the time from randomization to the first documented PD per RECIST 1.1 based on assessments by investigator or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Objective response rate (ORR) assessed by BIRC or investigators | Up to approximately 37 months from first patient in
  ORR is defined as the percentage of participants in the analysis population who have a complete response (CR: disappearance of all lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experienced a CR or PR as assessed by BIRC or investigators based on RECIST 1.1 is presented.
Disease control rate (DCR) assessed by BIRC or investigators | Up to approximately 37 months from first patient in
  DCR is defined as the sum rate of CR, PR and Stable Disease (SD), as determined by BIRC or investigators using RECIST v1.1
Duration of response (DoR) assessed by BIRC or investigators | Up to approximately 37 months from first patient in
  DoR is defined as the time period from the date of initial CR or PR until the date of PD or death due to any cause, whichever occurs first.
Incidence and severity of Adverse Event (AE) according to CTCAE 5.0 | Up to 30 days after last treatment
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Differences in the scores of health-related quality of life (HRQol) evaluated by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) | Up to 30 days after last treatment
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" (Item 29) and "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores were standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score are presented.
Differences in the scores of health-related quality of life (HRQol) evaluated by EORTC Quality of Life Questionnaire - Breast Cancer (QLQ-BR42) | Up to 30 days after last treatment
  Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score denotes worse symptoms for the systemic therapy side effects symptom scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, professor, Study Chair — Fudan University; Jian Zhang, professor, Study Chair — Fudan University
Locations (70):
- China (70):
  - The first affiliated hospital of bengbu medical University, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Southwest Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Lanzhou University First Hospital, Lanzhou, Gansu
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Affillated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital Affiliated to Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Affiliated Anyang Tumor Hospital of Henan University of Science and Technology, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital Tongji Medical College of Hust, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangyang Cancer Hospital, Xiangyang, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - The Second Hospital Of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Ruijin hospital of Shanghai Jiao Tong university School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi cancer hospital, Taiyuan, Shanxi
  - Runcheng City Center Hospital, Yuncheng, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Nanchong Central Hospital of Sichuan Province, Nanchong, Sichuan
  - The First People's Hospital of Neijiang, Neijiang, Sichuan
  - The Second People's Hospital Of Neijiang, Neijiang, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tian Jin Medicial University Cancer Institute&Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital (The Third Affiliated Hospital of Kunming Medical University), Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract,articles or papers) or any presentations.
Time Frame: After the trial completed
Access Criteria: NCI is committed to sharing data in accordance with NIH policy